CLINICAL TRIAL: NCT04533607
Title: Modular Approach for Autism Programs in Schools
Acronym: MAAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: May Institute (Other)
Collaborators: University of South Florida (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Cynthia Anderson, Senior Vice President of Applied Behavior Analysis and Director of the National Autism Center, May Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R324A200154
Record Dates: First submitted 2020-08-20; First posted 2020-08-31 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; autism; ASD
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Schools will be randomized to either MAAPS or waitlist control with equal probability. Randomization at the school level will minimize the risk of spillover between MAAPS and the waitlist control group. Randomization will be conducted for each site to guarantee equal representation of treatment and control schools at each site. The project statistician will generate a randomization sequence that is concealed from the study team.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAAPS (Active Comparator): Modular intervention system integrating evidence-based strategies to address core and associated features of ASD and ongoing coaching.
  Interventions: Behavioral: MAAPS
- Waitlist control (No Intervention): Services as usual.

INTERVENTIONS:
Behavioral: MAAPS — Modular intervention system integrating evidence-based strategies to address core and associated features of ASD and ongoing coaching.
  Arms: MAAPS

SUMMARY:
The number of students aged 6-21 years with an educational classification of autism spectrum disorder (ASD) in the United States grew by about 19 times over a 19-year period-from 29,076 in 1995-6 to 545,198 in 2014-2015 (IDEA Data Center, 2018). Meeting the needs of this growing population of students is a significant concern for schools (Bowen, 2014). Investigators have described as many as 27 efficacious intervention strategies for teaching new skills to children with ASD (Wong et al., 2015). However, these strategies are only rarely implemented in schools. In a survey of 185 teachers across the state of Georgia working with at least one student with ASD, fewer than 5% reported using an evidence-based intervention (Hess, Morrier, Heflin, & Ivey, 2008). To address gaps in current practice for students with ASD, there is a need for (1) a process for selecting and implementing interventions that can address the multi-faceted needs of students with ASD and (2) a service-delivery system that is feasible, flexible, durable, effective, and sustainable in schools. The investigators hypothesize that The Modular Approach for Autism Programs in Schools (MAAPS), an individualized, comprehensive modular intervention system, will address this gap. MAAPS integrates evidence-based strategies to address core and associated features of autism spectrum disorders (ASD) to enhance the success of elementary students with ASD in schools. The primary aim is to evaluate whether, compared to services as usual, MAAPS improves teacher outcomes and subsequent student educational outcomes.

DETAILED DESCRIPTION:
Background: The number of students aged 6-21 years with an educational classification of autism spectrum disorder (ASD) in the United States grew by about 19 times over a 19-year period-from 29,076 in 1995-6 to 545,198 in 2014-2015 (IDEA Data Center, 2018). Meeting the needs of this growing population of students is a significant concern for schools (Bowen, 2014). Investigators have described as many as 27 efficacious intervention strategies for teaching new skills to children with ASD (Wong et al., 2015). However, these strategies are only rarely implemented in schools. In a survey of 185 teachers across the state of Georgia working with at least one student with ASD, fewer than 5% reported using an evidence-based intervention (Hess, Morrier, Heflin, & Ivey, 2008). The infrequent use of the wide range of evidence-based strategies that could improve outcomes for students with ASD is concerning and may at least partially explain why students with ASD receive large amounts of special education services (Brookman-Frazee et al., 2009) yet often continue to require extensive supports as adults (Howlin et al., 2004).

Objectives: The purpose of this project is to test the efficacy of the Modular Approach for Autism Programs in Schools (MAAPS). The Modular Approach for Autism Programs in Schools (MAAPS) is an individualized, comprehensive modular intervention system integrating evidence-based strategies to address core and associated features of autism spectrum disorders (ASD) to enhance the success of elementary students with ASD in schools.

Specific Aims: The primary aim is to evaluate whether, compared to services as usual, MAAPS improves teacher outcomes and subsequent student educational outcomes. The investigators also intend to explore the feasibility and acceptability of MAAPS, costs associated with MAAPS, and analyze any potential modifiers of intervention effects and the implementation process.

Design: 60 schools will be randomized to either MAAPS or waitlist control. 120 teacher-student dyads will be enrolled from these 60 schools. Schools will be recruited from three sites: May Institute, University of South Florida, and University of Rochester. Student outcome measures assess overall school functioning, improvements in teacher-nominated target behaviors, core and associated features of ASD. Teacher outcome measures assess feasibility, acceptability, and usability of MAAPS and teacher implementation fidelity.

ELIGIBILITY:
Inclusion Criteria:

* Educational classification of autism spectrum disorder
* Attending a public elementary school (K-6th grade)
* Attending school in person at least one day per week
* No planned changes in school placement or core team members in upcoming school year
* Parents/guardians able to participate in study-related activities (e.g., informed consent process and completion of study measures)
* Child's teacher consents to participate

Exclusion Criteria:

* Profound vision or hearing loss
* Motor disabilities such as cerebral palsy
* Genetic disorder known to be associated with ASD such as Fragile X, Down Syndrome, tuberous sclerosis

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in score for Developmental Disability-Clinical Global Assessment Scale (DD-CGAS) | Baseline, approximately 6 months after baseline, approximately 9 months after baseline
  This measure will be used to assess overall functioning. The DD-CGAS is a rating scale with scores from 1 (extreme and pervasive impairment) to 100 (superior functioning).
Change in rating for Teacher Nominated Target Problems (TNTP) | Baseline, approximately 6 months after baseline, approximately 9 months after baseline
  This measure represents the three most pressing, operationalized target problems for each student. Target problems are specified with specific descriptions of intensity/frequency at baseline. Following baseline, ratings of improvement are gathered for each target problem on a 7-point Likert scale, ranging from 1= very much improved, good functioning, minimal symptoms, substantial change to 7= very much worse, severe exacerbation of symptoms and loss of functioning.
Change in score for Social Skills Improvement System (SSIS) | Baseline, approximately 6 months after baseline, approximately 9 months after baseline
  This measure will be used to assess social communication and interaction and problem behavior and will be completed by the teacher. The SSIS has several subscales that use a 4-point Likert scale to rate the frequency of specified behaviors and a 3-point Likert rating the importance of each item. The 30-item Social Skills Subscale is a measure of social communication and interaction. The SSIS Problem Behaviors Scale will be used to assess problem behavior. This scale includes 18 items that can be interpreted independently of the SSIS composite score. This will be administered for students emitting challenging behavior.
Change in score for Children's Communication Checklist, Second Edition (CCC-2) | Baseline and approximately 9 months after baseline
  The CCC-2 is a 5-10-minute rating scale that assesses communication skills in the areas of pragmatic language, syntax, word formation, semantics, and overall speech. It yields an index that includes clinical cutoffs to indicate profiles consistent with ASD.
Change in score for Children's Yale-Brown Obsessive-Compulsive Scales-ASD (CYBOCS-ASD) | Baseline, approximately 6 months after baseline, approximately 9 months after baseline
  This measure will be used to assess restricted and repetitive behavior. The CYBOCS-ASD is a semi-structured clinician-rated scale designed to rate the current severity of repetitive behavior in children with ASD. A five-point Likert scale is used for rating with a 0 indicating less symptomatic to a 4 indicating most symptomatic. A total score is obtained ranging from 0-20.
Change in engaged time measured by Academic Engaged Time (AET) | Baseline, approximately 6 months after baseline, approximately 9 months after baseline
  This measure will be used to assess academic functioning. An independent data collector directly observes the student for two 15-minute instructional periods. A stopwatch is used to record the duration of time the student is preforming engaged behaviors. Two observations will be administered at the relevant timepoints.
Change in score for Adaptive Behavior Assessment System, Third Edition (ABAS-3) | Baseline and approximately 9 months after baseline
  The raw score from the 21-item Self Direction Scale will be used to measure school-related adaptive functioning. This subscale is a nationally normed, well-established, 15-minute questionnaire measuring school-related adaptive functioning. It is validated to use independent of the ABAS-3 total score.

SECONDARY OUTCOMES:
Usage Rating Profile-Intervention, Revised (URP-IR) | Approximately 9 months after baseline
  This measure will be used to measure social validity. The URP is a 29-item, 6-point rating scale with six factors: acceptability, understanding the intervention, home-school collaboration needed, feasibility, system climate and systems support needed for the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Anderson, PhD, BCBA-D-D, Principal Investigator — May Institute
Locations (3):
- United States (3):
  - University of South Florida, Tampa, Florida
  - Kaitlin M Gould, Randolph, Massachusetts
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: No